CLINICAL TRIAL: NCT02420873
Title: An Open-label Phase II Study of Lorvotuzumab Mertansine (IMGN901) in CD56 Expressing Hematological Malignancies
Brief Title: An Open-label Phase II Study of Lorvotuzumab Mertansine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: ImmunoGen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0926; NCI-2015-00683 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Results first posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Leukemia
Keywords: Leukemia; Hematological malignancy; Myelofibrosis; MF; Blastic plasmacytoid dendritic cell neoplasm; BPDCN; CD56 tumor marker; Acute myeloid leukemia; AML; Natural-killer leukemia; Acute lymphoblastic leukemia; ALL; CD56 expressing hematological malignancy; IMGN901; Lorvotuzumab mertansine
MeSH Terms: conditions — Leukemia; Hematologic Neoplasms; Primary Myelofibrosis; Blastic Plasmacytoid Dendritic Cell Neoplasm; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — lorvotuzumab mertansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: CD56 Expressing Hematological Malignancies (Experimental): Lorvotuzumab mertansine (IMGN901) administered intravenously at a dose of 100 mg/m2 on Day 1 and 8 of a 21-day cycle.
  Interventions: Drug: Lorvotuzumab Mertansine (IMGN901)
- Cohort 2: Myelofibrosis (Experimental): Lorvotuzumab mertansine (IMGN901) administered intravenously at a dose of 100 mg/m2 on Day 1 and 8 of a 21-day cycle.
  Interventions: Drug: Lorvotuzumab Mertansine (IMGN901)
- Cohort 3: Blastic Plasmacytoid Dendritic Cell Neoplasm (Experimental): Lorvotuzumab mertansine (IMGN901) administered intravenously at a dose of 100 mg/m2 on Day 1 and 8 of a 21-day cycle.
  Interventions: Drug: Lorvotuzumab Mertansine (IMGN901)

INTERVENTIONS:
Drug: Lorvotuzumab Mertansine (IMGN901) — 100 mg/m2 by vein on Day 1 and 8 of a 21-day cycle.

SUMMARY:
The goal of this clinical research study is to learn if lorvotuzumab mertansine can help to control blood cancers that have the CD56 tumor marker. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
Study Treatment:

If you are found to be eligible to take part in this study, you will receive lorvotuzumab by vein on Days 1 and 8 (+/- 2 days) of each cycle. It may take a few minutes or several hours to receive the study drug. Your doctor will discuss this with you.

All treatments with IMGN901 must be administered at MD Anderson.

Each cycle is 21 days (+/-6 days). However, they may be longer or shorter depending on if/how the disease responds to the treatment, how your bone marrow reacts to treatment, and what the doctor thinks is in your best interest.

Your dose of lorvotuzumab may be raised, lowered, and/or delayed if the doctor thinks it is in your best interest.

Study Visits:

On Day 1 of each cycle, you will have a physical exam.

One (1) time each week during the first 4 cycles, blood (about 1 tablespoon) will be drawn for routine tests. After Cycle 4, you will have these blood draws 1 time every 2-4 weeks. If your doctor thinks it is needed, more blood may need to be drawn. The study doctor or study staff will discuss this with you if more blood is needed.

During the first cycle, all the laboratory evaluations will be done at MD Anderson. After Cycle 1, you may be able to have these blood draws performed at a local lab or clinic that is closer to your home, and the results reported to the research nurse of the study at MD Anderson. The study doctor or study staff will discuss this option with you. The results of these blood draws will be sent to the study doctor for review.

On Day 21 of Cycle 1 (+/- 7 days), then every 1-3 cycles after that, you will have a bone marrow aspiration/biopsy to check the status of the disease. If the doctor thinks it is needed, these may be done more or less often, depending on your response to the study drug.

You will have blood draws and/or bone marrow aspirations at any time that the doctor thinks it is needed while you are on study.

If you stay on study for more than 6 months and you are not having side effects, you may have some of the above tests more or less frequently. For example, you may only have a bone marrow aspiration 1 time every 6-12 months and blood draws 1 time each cycle. The study doctor will discuss this with you.

Length of Study:

You may take up to 12 cycles of lorvotuzumab. If the doctor thinks it is in your best interest, you may be able to continue receiving the study drug beyond Cycle 12. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after follow-up.

End-of-Study Visit:

If you leave the study before the end of Cycle 12, within 30 days (+/- 7 days) after the last dose of study drug:

* Blood (about 2-3 tablespoons) will be drawn for routine tests.
* If the doctor thinks it is needed, you will have a bone marrow aspirate/biopsy to check the status of the disease.

Long Term Follow-Up:

If the disease appears to get better and you are responding well to the study drug, you will return to MD Anderson every 3-6 months for up to 5 years after your last dose of study drug for the study staff to check how you are doing.

If you cannot return to MD Anderson for these visits, you may be called by a member of the study staff. The call should last about 10 minutes.

This is an investigational study. Lorvotuzumab is not FDA approved or commercially available. It is currently being used for research purposes only. The study doctor can explain how the drug is designed to work.

Up to 60 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CD56 expressing hematological malignancy, as follows: Cohort 1: CD56 expressing hematological malignancies including but not limited to AML, high-risk myelodysplastic syndrome (MDS), natural-killer leukemia, acute lymphoblastic leukemia, accelerated and blast-phase chronic myelocytic leukemia (CML) who have failed prior therapy or for which no standard therapy exists.Cohort 2: Patients with MF (either primary MF, post-polycythemia MF, or post-essential thrombocythemia MF) and CD56 expression who have been on ruxolitinib or JAK-inhibitor therapy for at least 12 weeks and deemed refractory or sub-optimal responders in the opinion of the treating physician.Cohort 3: Patients with pathological diagnosis of BPDCN with CD56 expression (frontline and relapsed/refractory).
2. Any level of CD56 expression will be considered sufficient for enrollment on this study.
3. Prior therapy with hydroxyurea, chemotherapy, biological or targeted therapy (e.g. FLT3 inhibitors, other kinase inhibitors), or hematopoietic growth factors is allowed.
4. Age >/=18 years
5. Eastern Cooperative Oncology Group (ECOG) Performance Status </= 2
6. Adequate organ function: total bilirubin </= 2 times upper limit of normal (x ULN) (</=3 x ULN if considered to be due to leukemic involvement or Gilbert's syndrome); aspartate aminotransferase (AST) or alanine aminotransferase (ALT) </= 2.5 x ULN (</= 5.0 x ULN if considered to be due to leukemic involvement); serum creatinine </= 2 x ULN, amylase and lipase </=2 x ULN .
7. In the absence of rapidly progressing disease and after discussion with the Principal Investigator (PI), the interval from prior treatment to time of IMGN901 administration will be at least 2 weeks or at least 5 half-lives for cytotoxic/noncytotoxic agents. The half-life be based on published pharmacokinetic literature (abstracts, manuscripts, investigator brochure's, or drug-administration manuals) and will be documented in the protocol eligibility document.
8. continuation from criteria #7: For prior monoclonal antibody therapy the interval from prior monoclonal antibody treatment to time of IMGN901 administration will be at least 2 weeks. The use of chemotherapeutic or anti-leukemic agents other than hydroxyurea (as defined in the protocol) is not permitted during the study with the exception of intrathecal (IT) therapy for patients with controlled CNS leukemia at the discretion of the PI. Hydroxyurea is allowed prior to the initiation of IMGN901 and during the first 3 cycles, either prior to or concomitantly with IMGN901 administration initially to control Leukocytosis.
9. Women of childbearing potential must practice contraception. Females of childbearing potential: Recommendation is for 2 effective contraceptive methods during the study. Adequate forms of contraception are double barrier methods (condoms with spermicidal jelly or foam and diaphragm with spermicidal jelly or foam), oral, depo provera, or injectable contraceptives, intrauterine devices, and tubal ligation. Male patients with female partners who are of childbearing potential: Recommendation is for male and partner to use at least 2 effective contraceptive methods, as described above, during the study.
10. Females must be surgically or biologically sterile or postmenopausal (amenorrheic for at least 12 months) or if of childbearing potential, must have a negative serum or urine pregnancy test within 72 hours before the start of the treatment
11. Patients must provide written informed consent.
12. Women of childbearing potential must agree to use an adequate method of contraception during the study and until 3 months after the last treatment. Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study until 3 months after the last treatment. Adequate methods of contraception include: Total abstinence when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment Male sterilization (at least 6 months prior to screening).
13. continued from criteria #12: For female patients on the study, the vasectomized male partner should be the sole partner for that patient Combination of any of the two following (a+b or a+c or b+c) Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception Placement of an intrauterine device (IUD) or intrauterine system (IUS) Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository In case of use of oral contraception, women should have been stable on the same pill before taking study treatment. Note: Oral contraceptives are allowed but should be used in conjunction with a barrier method of contraception due to unknown effect of drug-drug interaction
14. continued from criteria #13 Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.

Exclusion Criteria:

1. Patients with known allergy or hypersensitivity to IMGN901.
2. Patients who have previously been treated with IMGN901.
3. Patients with symptomatic central nervous system (CNS) leukemia or patients with poorly controlled central nervous system leukemia.
4. Peripheral neuropathy >grade 2.
5. Active or clinically symptomatic chronic pancreatitis or disease affecting pancreas.
6. Neurologic disease including multiple sclerosis, Eaton-Lambert syndrome, demyelination.
7. Significant cardiac disease including myocardial infarction or unstable angina within 6 months, uncontrolled hypertension despite medical therapy (defined as blood pressure >160/110 in spite of adequate medical therapy), active and uncontrolled congestive heart failure New York Heart Association (NYHA) class III/IV, stroke within preceding 6 months.
8. Patients with known Human Immunodeficiency Virus seropositivity will be excluded.
9. Known to be positive for hepatitis B by surface antigen expression. Known to have active hepatitis C infection (positive by polymerase chain reaction or on antiviral therapy for hepatitis C within the last 6 months). Known to be active CMV infection or herpes zoster infection.
10. Pregnant or breast feeding (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive B-human chorionic gonadotropin (HCG) laboratory test.
11. Patients with any concurrent severe and/or uncontrolled medical condition or active uncontrolled systemic infection as determined by the investigator.
12. Patients who have had any major surgical procedure within 14 days of Day 1.
13. Patients unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-05-12 (Actual); Primary Completion 2017-06-06 (Actual); Study Completion 2017-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naval Daver, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: May 2015 through July 2016. All of the participants were recruited at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: All of the participants registered on this study have CD56 expressing hematological malignancies and were assigned to cohort 1 of this study. No participants registered on this study had a diagnosis of Myelofibrosis or Blastic Plasmacytoid Dendritic Cell Neoplasms, Therefore, zero participants were analyzed on cohort 2 or cohort 3 of this study.
Period: Overall Study
Arm/Group | Cohort 1: CD56 Expressing Hematological Malignancies | Cohort 2: Myelofibrosis | Cohort 3: Blastic Plasmacytoid Dendritic Cell Neoplasm
Started | 9 | 0 | 0
Completed | 9 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Zero participants were registered on Cohort 2 (Myelofibrosis arm) or Cohort 3 (Blastic Plasmacytoid Dendritic Cell Neoplasm arm).
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: CD56 Expressing Hematological Malignancies | Cohort 2: Myelofibrosis | Cohort 3: Blastic Plasmacytoid Dendritic Cell Neoplasm | Total
Number analyzed (Participants) | 9 | 0 | 0 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 0 | 0 | 8
  >=65 years | 1 | 0 | 0 | 1
Age, Continuous [Median (Full Range); unit: years] | 58 [28 to 72] |  |  | 58 [28 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 0 | 5
  Male | 4 | 0 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 7 | 0 | 0 | 7
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 |  |  | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) of IMGN901 in Participants CD56 Expressing Hematological Malignancies
Description: ORR, defined as CR (complete remission) + CRp (complete remission with incomplete platelet recovery) + CRi (complete remission with incomplete count recovery) within 3 cycles of therapy with IMGN901.
Time Frame: 53 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: CD56 Expressing Hematological Malignancies | Cohort 2: Myelofibrosis | Cohort 3: Blastic Plasmacytoid Dendritic Cell Neoplasm
Number analyzed (Participants) | 9 | 0 | 0
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events reported during each treatment course. Overall period: May 2015 to April 2016.
Description: Zero participants were registered on Cohort 2 (Myelofibrosis arm) or Cohort 3 (Blastic Plasmacytoid Dendritic Cell Neoplasm arm).
Arm/Group | Cohort 1: CD56 Expressing Hematological Malignancies | Cohort 2: Myelofibrosis | Cohort 3: Blastic Plasmacytoid Dendritic Cell Neoplasm
All-Cause Mortality (participants affected / at risk) | 4/9 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 9/9 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 6/9 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: CD56 Expressing Hematological Malignancies (N=9) | Cohort 2: Myelofibrosis (N=0) | Cohort 3: Blastic Plasmacytoid Dendritic Cell Neoplasm (N=0)
Abdominal Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Febrile Neutropenia (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Lung Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Multi-Organ Failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vulval Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: CD56 Expressing Hematological Malignancies (N=9) | Cohort 2: Myelofibrosis (N=0) | Cohort 3: Blastic Plasmacytoid Dendritic Cell Neoplasm (N=0)
Abdominal Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile Neutropenia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis Leg (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Increased Alanine Aminotransferase (ALT) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Anxiety (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Aspartate Aminotransferase (AST) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bone Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Cough (General disorders) | 2 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Ear Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Edema Limbs (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 2 (2) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophosphatemia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Hypoxia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
numbness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathy (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2015-07-16): https://cdn.clinicaltrials.gov/large-docs/73/NCT02420873/Prot_000.pdf
  • Statistical Analysis Plan (2015-07-16): https://cdn.clinicaltrials.gov/large-docs/73/NCT02420873/SAP_001.pdf